CLINICAL TRIAL: NCT01695837
Title: Live Well: A Practical and Effective Low-Intensity Dietary Counseling Intervention for Use in Primary Care Patients With Dyslipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Doina Kulick, MD, Associate Professor of Medicine, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5P20RR016464-11/8; 5P20RR016464 (NIH)
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Dyslipidemia
Keywords: Diet counseling; primary care
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A-dietary counseling month 0-6 (Experimental): Group A Visit #1 - Weight, height, blood pressure and pulse were measured at the beginning of the visit. During a "focused office visit" the primary care physician (PCP) reviewed the results of the fasting lipid panel and diet test with the patient; the PCP provide the patient with written educational materials and access to the counseling website. Weekly automatic emails sent to patient reminding to visit the counseling website
  Visit #2 - Same as visit #1. Weekly automatic emails sent to patient reminding to visit the counseling website.
  Visit #3 - Weight, blood pressure and pulse were measured at the beginning of the visit. During a "focused office visit" the PCP reviewed the results of the new fasting lipid panel and diet test with the patient.
  Interventions: Behavioral: Group A: Dietary counseling month 0-6 Group B: Dietary counseling month 3-6
- Group B- Dietary counseling month 3-6 (Other): Group B Visit #1: Weight, height, blood pressure and pulse were measured at the beginning of the visit. Follow up visit and lab order were scheduled for 3 months. No blood test or diet test results were reviewed with the patient.
  Visit #2 - Weight, blood pressure and pulse were measured at the beginning of the visit. During a "focused office visit" the PCP reviewed the results of the two fasting lipid panels ; the PCP provide the patient with written educational materials and access to the counseling website. Weekly automatic emails sent to patient reminding to visit the counseling website
  Visit #3 - Weight, blood pressure and pulse were measured at the beginning of the visit. During a "focused office visit" the PCP reviewed the results of the new fasting lipid panel and diet test with the patient.
  Interventions: Behavioral: Group A: Dietary counseling month 0-6 Group B: Dietary counseling month 3-6

INTERVENTIONS:
Behavioral: Group A: Dietary counseling month 0-6 Group B: Dietary counseling month 3-6

SUMMARY:
The purpose of this study was to evaluate the effects on lipids and diet of a low-intensity dietary counseling intervention provided by the primary care physician (PCP), in patients at risk for cardiovascular diseases

DETAILED DESCRIPTION:
The objective of this study is to design and evaluate the feasibility and the effect on diet quality and blood lipids a new dietary counseling intervention that will be sustainable in the "real-world" settings of the current clinical practice. The intervention will be initiated by the primary care physician during the routine office visits and will use paper and web-based counseling materials. Internet based healthcare, or e-healthcare, is a consumer focused health care delivery paradigm that physicians and the healthcare system can no longer ignore. Lifestyle counseling and preventive medicine are potentially ideal areas of patient care that could be provided efficiently through this emerging venue of healthcare delivery. Internet access is near-universal for Americans under the age of 60: 90% of 18-29 year-olds, 85% of 30-49 year-olds, and 70% of 50-64 year-olds.

The aims of this study are: 1) - develop a patient self-administered, computerized version of the paper-based Rate-your-Plate dietary screening Questionnaire; 2) - create counseling materials on diet and cholesterol and build a secure, HIPAA compliant, interactive web-based counseling application that will allow patients to receive personalized counseling base on the results of the screening dietary questionnaire and the goals chosen by the patients; 3) - to test the feasibility of this intervention in the clinical settings of primary care, and evaluate its effect on lipids panel at 3 and 6 months .

ELIGIBILITY:
Inclusion Criteria:

* Eligibility required documentation of a LDL-cholesterol level of 130 mg/dL or higher within the 12 months prior to enrollment. Potential subjects were also required to have access to the Internet and an active email account. The use of lipid lowering drugs was not an exclusion, but patients taking these drugs had be on the same medication and dose for at least 3 months prior to enrollment, with no changes anticipated for the duration of the trial.

Exclusion Criteria:

* We excluded patients with poorly controlled diabetes mellitus (defined by HbA1c>9%), serum creatinine above 1.5 mg/dL, malignancy, cirrhosis, eating disorders, acute coronary syndrome in the last three months, congestive heart failure NYHA class lll and lV, ongoing warfarin therapy, uncontrolled hypo- or hyperthyroidism, ongoing weight loss, history of bariatric surgery, pregnant women, and patients who scored more than 250 (on a scale of 100 to 300) on a food frequency questionnaire administered on the day of enrollment. Patients with a history of triglycerides >400 mg/dl were also excluded, since we used the Friedewald formula [LDL-C=Total cholesterol-(TGs/5+HDL-C)] to calculate LDL-cholesterol levels.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
LDL-Cholesterol | up to 6 months

SECONDARY OUTCOMES:
Total Cholesterol | at 3 and 6 months
Triglycerides | at 3 and 6 months
HDL-Cholesterol | at 3 and 6 months
diet score | at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Doina Kulick, MD, MS, Study Director — University of Nevada School of Medicine
Locations (1):
- UNSOM Internal Medicine, Reno, Nevada, United States

REFERENCES:
- [Derived] Kulick D, Langer RD, Ashley JM, Gans KM, Schlauch K, Feller C. Live well: a practical and effective low-intensity dietary counseling intervention for use in primary care patients with dyslipidemia--a randomized controlled pilot trial. BMC Fam Pract. 2013 May 12;14:59. doi: 10.1186/1471-2296-14-59. PMID 23663789